CLINICAL TRIAL: NCT03415945
Title: Left Ventricular Septal Pacing: Potential Application for Cardiac Resynchronization Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL58809.068.16
Record Dates: First submitted 2017-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy; Left Bundle-Branch Block
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRT implantation (Experimental): In cardiac resynchronization therapy (CRT), biventricular pacing is performed by pacing the right ventricle (RV) and epicardium of the left ventricular (LV) posterolateral wall.
  Interventions: Device: Cardiac resynchronization therapy (CRT)

INTERVENTIONS:
Device: Cardiac resynchronization therapy (CRT) — All study participants have a clinical indication for CRT and will receive CRT implantation as part of their routine medical care. Additionally, participants will receive temporary left and right ventricular septal pacing electrodes and a temporary PressureWire to investigate the acute hemodynamic effect of left ventricular septal pacing, using patients as their own controls.

SUMMARY:
In cardiac resynchronization therapy (CRT), biventricular pacing is performed by pacing the right ventricle (RV) and epicardium of the left ventricular (LV) postero-lateral wall. A significant proportion of apparently suitable patients fail to benefit from CRT. One of the problems of CRT is proper positioning and fixation of the LV pacing lead in the coronary vein. LV septal pacing may be a good alternative for BiV pacing in patients with an indication for CRT.

DETAILED DESCRIPTION:
Cardiac pump function depends on physiological electrical activation of the ventricles. This normal activation is disturbed during artificial electrical stimulation (pacing) of the right ventricle (RV), the common therapy to treat symptomatic slow heart rate ("rate control"), as well as during electrical dyssynchrony such as left bundle branch block (LBBB). As a consequence, RV pacing and LBBB reduce cardiac pump function and increase cardiac morbidity and mortality. During the last two decades cardiac resynchronization therapy (CRT) has emerged as treatment to "resynchronize" ventricular electrical activation by pacing the RV apical septum and left ventricular (LV) postero-lateral wall simultaneously ("biventricular" (BiV) pacing).

Since initial approval of the therapy over 10 years ago, there have been hundreds of thousands of implants performed worldwide. In the Netherlands currently more than 2000 CRT devices are implanted each year. Large clinical trials have shown that CRT improves LV systolic pump function, reverses structural remodelling, improves quality of life and exercise tolerance, and decrease mortality. However, a significant proportion of apparently suitable patients fail to benefit. Depending on the definition used, the response to CRT is positive in 50-70% of treated patients, leaving 30-50% without significant effect. One of the problems of CRT is proper positioning and fixation of the LV pacing lead in the coronary vein.

Research in the laboratory of the the investigators revealed that in dogs with AV-block and in patients with sinus node disease, pacing at the LV endocardial side of the interventricular septum (LV septal pacing) provides near physiological ventricular activation, near uniform distribution of workload, and near normal pump function. Furthermore, pump function during LV septal pacing was at least as good as during BiV pacing. A recent study, with acute hemodynamic data in dogs with LBBB and in a small group of patients with LBBB, further indicates that LV septal pacing may be used for CRT. A weakness of the patient data is that these patients were either non-responders to conventional CRT or patients where no access to the coronary sinus was obtained. Therefore, this group may not be representative for the entire CRT candidate population.

Two factors appear to determine the positive effect of LV septal pacing: the slow impulse conduction across the interventricular septum and the fast impulse conduction along the inner layers of the LV wall through superficial, non-Purkinje fibers. Following this reasoning, the investigators expect that the exact pacing site at the septum is not critical. This would be of great advantage for future applications in patients, since proper implantation of an LV lead in the coronary sinus requires attention in order to position the lead in the latest activated region.

The aim of the present study is to compare the electrophysiological and hemodynamic effects of several modes and sites of LV septal pacing with those of BiV pacing in patients undergoing CRT device implantation. The results may have a large impact on future pacing therapy. The LV septum may become an alternative for BiV pacing, but easier to apply, less invasive, and more cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure with NYHA functional class II-IV
* Left ventricular ejection fraction (LVEF) < 35%
* LBBB and QRS duration ≥ 130 ms or non-LBBB and QRS duration ≥ 150 ms
* In sinus rhythm
* Optimal pharmacological therapy

Exclusion Criteria:

* Persistent atrial fibrillation
* ≥ 2 premature ventricular complexes on standard 12-lead electrocardiogram (ECG)
* Age < 18 years
* Incapable of giving informed consent
* Moderate to severe aortic valve stenosis
* Peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-05-23 (Estimated); Study Completion 2020-05-23 (Estimated)

PRIMARY OUTCOMES:
Acute hemodynamic effect (LV dP/dtmax) of the best LV septal pacing side and conventional BiV pacing. | The outcome measure will be assessed during the CRT implantation procedure (the total procedure time will increase 45 to 60 minutes).
  A RadiAnalyzer Physio monitor version 2.02 (St. Jude Medical, St. Paul, USA) is used to calculate LV dP/dtmax as a measure of LV systolic function.

SECONDARY OUTCOMES:
Acute hemodynamic effects (LV dP/dtmax) of the different LV septal pacing sides with RV apical septum pacing, His pacing, RV septum pacing, LV epicardial postero-lateral wall pacing and intrinsic ventricular activation. | The outcome measure will be assessed during the CRT implantation procedure (the total procedure time will increase 45 to 60 minutes).
  A RadiAnalyzer Physio monitor version 2.02 (St. Jude Medical, St. Paul, USA) is used to calculate LV dP/dtmax as a measure of LV systolic function.
The effect on the sequence of LV electrical activation and body surface electrocardiographic mapping | The outcome measure will be assessed during the CRT implantation procedure (the total procedure time will increase 45 to 60 minutes).
  The sequence of LV electrical activation will be assessed by 3-dimensional vectorcardiography (VCG) and non-invasive body surface electrocardiographic mapping using the Verathon Heartscape system (developed by Medtronic)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Vernooy, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Mills RW, Cornelussen RN, Mulligan LJ, Strik M, Rademakers LM, Skadsberg ND, van Hunnik A, Kuiper M, Lampert A, Delhaas T, Prinzen FW. Left ventricular septal and left ventricular apical pacing chronically maintain cardiac contractile coordination, pump function and efficiency. Circ Arrhythm Electrophysiol. 2009 Oct;2(5):571-9. doi: 10.1161/CIRCEP.109.882910. Epub 2009 Aug 25. PMID 19843926
- [Background] Mafi-Rad M, Luermans JG, Blaauw Y, Janssen M, Crijns HJ, Prinzen FW, Vernooy K. Feasibility and Acute Hemodynamic Effect of Left Ventricular Septal Pacing by Transvenous Approach Through the Interventricular Septum. Circ Arrhythm Electrophysiol. 2016 Mar;9(3):e003344. doi: 10.1161/CIRCEP.115.003344. PMID 26888445
- [Background] Strik M, Rademakers LM, van Deursen CJ, van Hunnik A, Kuiper M, Klersy C, Auricchio A, Prinzen FW. Endocardial left ventricular pacing improves cardiac resynchronization therapy in chronic asynchronous infarction and heart failure models. Circ Arrhythm Electrophysiol. 2012 Feb;5(1):191-200. doi: 10.1161/CIRCEP.111.965814. Epub 2011 Nov 7. PMID 22062796
- [Background] Strik M, van Deursen CJ, van Middendorp LB, van Hunnik A, Kuiper M, Auricchio A, Prinzen FW. Transseptal conduction as an important determinant for cardiac resynchronization therapy, as revealed by extensive electrical mapping in the dyssynchronous canine heart. Circ Arrhythm Electrophysiol. 2013 Aug;6(4):682-9. doi: 10.1161/CIRCEP.111.000028. Epub 2013 Jul 19. PMID 23873141
- [Background] Singh JP, Fan D, Heist EK, Alabiad CR, Taub C, Reddy V, Mansour M, Picard MH, Ruskin JN, Mela T. Left ventricular lead electrical delay predicts response to cardiac resynchronization therapy. Heart Rhythm. 2006 Nov;3(11):1285-92. doi: 10.1016/j.hrthm.2006.07.034. Epub 2006 Aug 10. PMID 17074633
- [Background] Kors JA, van Herpen G, Sittig AC, van Bemmel JH. Reconstruction of the Frank vectorcardiogram from standard electrocardiographic leads: diagnostic comparison of different methods. Eur Heart J. 1990 Dec;11(12):1083-92. doi: 10.1093/oxfordjournals.eurheartj.a059647. PMID 2292255
- [Background] Man S, Algra AM, Schreurs CA, Borleffs CJ, Scherptong RW, van Erven L, van der Wall EE, Cannegieter SC, Schalij MJ, Swenne CA. Influence of the vectorcardiogram synthesis matrix on the power of the electrocardiogram-derived spatial QRS-T angle to predict arrhythmias in patients with ischemic heart disease and systolic left ventricular dysfunction. J Electrocardiol. 2011 Jul-Aug;44(4):410-5. doi: 10.1016/j.jelectrocard.2011.04.007. PMID 21704219
- [Background] Schreurs CA, Algra AM, Man SC, Cannegieter SC, van der Wall EE, Schalij MJ, Kors JA, Swenne CA. The spatial QRS-T angle in the Frank vectorcardiogram: accuracy of estimates derived from the 12-lead electrocardiogram. J Electrocardiol. 2010 Jul-Aug;43(4):294-301. doi: 10.1016/j.jelectrocard.2010.03.009. Epub 2010 Apr 24. PMID 20417936